CLINICAL TRIAL: NCT03349736
Title: Pelvic Floor Muscle Training Programme in Pregnant Nepalese Women- a Feasibility Study
Acronym: PFMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kathmandu University School of Medical Sciences (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Ranjeeta Shijagurumayum Acharya, Physiotherapists,PT,MSc, Kathmandu University School of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 112/2016
Record Dates: First submitted 2017-11-05; First posted 2017-11-22 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Pelvic Organ Prolapse; Urinary Incontinence
Keywords: Pelvic floor muscle
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: A feasibility study including 250 women to assess the feasibility of performing PFMT in pregnant Nepalese women. The PFMT programme consisted of attending a minimum of four supervised PFMT follow-up visits after inclusion to the programme and to perform PFMT daily at home.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pelvic Floor Muscle Training (Other): Women visiting antenatal (up to16 weeks of gestation) will be enrolled for the study. The women will be follow up 4 times during the antenatal visit until 37 weeks of gestation. Questionnaire data and clinical measurements(strength of PFM by Electromyograph biofeedback) will be registered at baseline and and follow-up at week 37 of pregnancy.
  The treatment program will include
  1) Information, educational material (leaflets, posters, and video) and individual/group exercise on PFM exercise on the 1st day of the visit. Counseling about the importance of performing PFM exercise will be provided. Women are advised to perform home PFM exercise and record in the exercise diary.
  Interventions: Other: Pelvic Floor Muscle Training

INTERVENTIONS:
Other: Pelvic Floor Muscle Training — All the women will receive information and instruction/guidance exercise individually and in groups on PFMT on the first day of their visit. Following this, the women are advised to perform daily PFMT at home which includes 10 sec hold X 10 times X 3 sets. Women will record their home PFMT using an exercise diary. During the follow-up, women will attend the PFMT in a group or individual led by a Physiotherapists (to motivate and to ensure women are performing the PFMT correctly). Exercise diary will be collected in every follow up so that the information is retained even if the women discontinued or deviate from intervention protocols.

SUMMARY:
To our knowledge, no studies in Nepal have reported the feasibility of performing the pelvic floor muscle training in Nepalese women. The aim of the study is to develop and a pelvic floor muscle training programme based on information, education (leaflet, video) and pelvic floor muscles (PFM) exercise in order to prevent or reduce Pelvic organ prolapse(POP) and Urinary Incontinence (UI) in pregnant Nepalese women.

The women will receive information (leaflet, video, posters) and guidance on PFMT. Following this, the women are advised to perform daily home PFM exercise Women will record their home PFMT using an exercise diary.

DETAILED DESCRIPTION:
PFM supports the bowel, bladder, and uterus. Pelvic floor dysfunction can lead to gynecological problems like POP and UI. POP is the downward displacement of uterus from its normal anatomical position and UI is the involuntary leakage of urine.

In Nepal, the prevalence of POP is 10% in women of reproductive age and reported UI is 60% and 50.6% from two studies. POP risk factors include early marriage, high parity, squatting during delivery, prolonged labor, increasing age, menopause, hysterectomy, smoking, obesity, heavy lifting, and early return to work after parturition. High reports of POP and UI could be due to the exposure to these potential risks factors in Nepalese women. Women in Nepal play a significant role in agricultural and household work and are exposed to these risks factors daily. Studies have shown that besides longer days with work, women have less time for sleep and leisure. One of the main work-related health problems for Nepalese women is the physical effect of chronic overwork due to women's triple roles and subordinate position in the family.

The government of Nepal created a fund to provide free surgery to women with POP in 2008. Surgery is a common treatment for POP, however, 58% report an occurrence of recurrent prolapse after surgery and 29% report re-operations. PFM exercise has Level I evidence for treatment (Stage 1 & 2) or prevention of POP. Women diagnosed with POP in Nepal, have 69.1% first-degree prolapse while the remaining 30.9% suffer from second and third-degree prolapse. Women's reluctance to seek treatment might be lack of family support, high costs for travel, food and lodging and ineffective treatment. Moreover, the health facilities are poor in rural areas as the infrastructure is weak, with few roads and commonly in poor condition which makes it more difficult. The PFM exercise does not need an instrument and can be done at home/workplace. PFM exercise for the treatment of POP (stage 1 & 2) and UI was popularized by Kegel exercise. The use of PFM exercise is based on two functions of the PFM, support of the pelvic organs and a contribution to the sphincter closure mechanism of the urethra.

This project will investigate the feasibility of a cost-effective physiotherapy program based on information, education, and PFMT, hopefully, to help improve the health outcome of Nepalese women. The feasibility study will be essential for a future cluster randomized controlled study.

Hence, the aim is to assess the feasibility of performing PFMT in pregnant women to help prevent or reduce POP and UI in Nepal.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women able to understand information and instructions in the Nepalese language

Exclusion Criteria:

* women with psychiatric diagnosis
* pregnancy related complications like pre-eclampsia
* risk of threatened abortion
* more than 16 weeks duration in 1st visit and
* not willing to participate or not able to communicate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study will be conducted in pregnant women
Enrollment: 253 (Actual)
Dates: Start 2017-06-25 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
To develop a PFMT programme and and second to assess the feasibility in terms of recruitment capability, sample characteristics, data collection procedures, outcome measures, and acceptability of the PFMT programme in pregnant Nepalese women. | 21 weeks
  Acceptability of the PFMT programme was assessed by attendance at supervised PFMT hospital visits, adherence to daily PFMT, and participant experiences of attending the programme.

CONTACTS AND LOCATIONS:
Overall Officials: Britt Stuge, PhD, Study Director — Oslo University Hospital; Rajendra Koju, MD, Study Chair — Kathmandu University School of Medical Sciences
Locations (1):
- Kathmandu University Dhulikhel Hospital, Kavre, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bo K, Frawley HC, Haylen BT, Abramov Y, Almeida FG, Berghmans B, Bortolini M, Dumoulin C, Gomes M, McClurg D, Meijlink J, Shelly E, Trabuco E, Walker C, Wells A. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for the conservative and nonpharmacological management of female pelvic floor dysfunction. Int Urogynecol J. 2017 Feb;28(2):191-213. doi: 10.1007/s00192-016-3123-4. Epub 2016 Dec 5. PMID 27921161
- [Background] Gurung G, Rana A, Amatya A, Bista KD, Joshi AB, Sayami J. Pelvic organ prolapse in rural Nepalese women of reproductive age groups:What makes it so common? Nepal Journal of Obstetrics and Gynaecology 2(2):35-41, 2007,
- [Background] Fitchett JR, Bhatta S, Sherpa TY, Malla BS, A Fitchett EJ, Samen A, Kristensen S. Non-surgical interventions for pelvic organ prolapse in rural Nepal: a prospective monitoring and evaluation study. JRSM Open. 2015 Nov 3;6(12):2054270415608117. doi: 10.1177/2054270415608117. eCollection 2015 Dec. PMID 26664731
- [Background] Regmi M, Uprety D, Poonam M. Prevalence of urinary incontinence among gynecological admissions at tertiary care hospital in eastern Nepal. Health Renaissance 10(1):16-9, 2012
- [Background] Pradhan A, Shrestha N. Working hour and its impact on backache from gender perspective. Dhaulagiri Journal of Sociology and Anthropology 4:235-46,2010
- [Background] Shrestha A, Lakhey B, Sharma J, Singh M, Shrestha B, Singh S. Prevalence of uterine prolapse amongst gynecology OPD patients in Tribhuwan university teaching hospital in Nepal and its socio-cultural determinants. Res Cent Women. 2009
- [Background] Hagen S, Stark D. Conservative prevention and management of pelvic organ prolapse in women. Cochrane Database Syst Rev. 2011 Dec 7;2011(12):CD003882. doi: 10.1002/14651858.CD003882.pub4. PMID 22161382
- [Background] Bodner-Adler B, Shrivastava C, Bodner K. Risk factors for uterine prolapse in Nepal. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Nov;18(11):1343-6. doi: 10.1007/s00192-007-0331-y. Epub 2007 Mar 1. PMID 17333434
- [Background] Shrestha B, Onta S, Choulagai B, Poudyal A, Pahari DP, Uprety A, Petzold M, Krettek A. Women's experiences and health care-seeking practices in relation to uterine prolapse in a hill district of Nepal. BMC Womens Health. 2014 Feb 3;14:20. doi: 10.1186/1472-6874-14-20. PMID 24490616
- [Background] Boyle R, Hay-Smith EJ, Cody JD, Morkved S. Pelvic floor muscle training for prevention and treatment of urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2012 Oct 17;10:CD007471. doi: 10.1002/14651858.CD007471.pub2. PMID 23076935
- [Background] KEGEL AH. Progressive resistance exercise in the functional restoration of the perineal muscles. Am J Obstet Gynecol. 1948 Aug;56(2):238-48. doi: 10.1016/0002-9378(48)90266-x. No abstract available. PMID 18877152